CLINICAL TRIAL: NCT01132924
Title: A Follow-up of the Early Pregnancy Study Cohort
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999910108; 10-E-N108
Record Dates: First submitted 2010-05-27; First posted 2010-05-28 (Estimated); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Gestational Age; Time to Pregnancy; Early Pregnancy Loss
Keywords: Early Pregnancy; Gestational Age; Fecundability; Ovulation; Recall; Natural History
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EPS Study Participants: Women who participated in the 1982-1986 North Carolina Early Pregnancy Study (EPS)

SUMMARY:
Background:

- The purpose of the 1982 1986 North Carolina Early Pregnancy Study was to determine how often pregnancy loss occurs before women know they are pregnant. Women planning to become pregnant were asked to collect daily urine specimens and fill out daily diaries of their intercourse and menstrual bleeding. Researchers are interested in re-contacting this cohort to gather new information and to examine how accurately women can recall events that occurred earlier in their lives.

Objectives:

- To follow-up with and gather additional information from women who were involved in the Early Pregnancy Study.

Eligibility:

- Women who participated in the 1982 1986 North Carolina Early Pregnancy Study.

Design:

* Participants will receive and complete a questionnaire that includes the following topics:
* Their pregnancy history.
* The infant s birth, including method of delivery and induction of labor.
* Early life exposures such as their own birth weight and their parents ages at their birth.
* Tap water use during their attempt to conceive
* General description of their behaviors during their participation in the original study, these include: physical activity, caffeine, alcohol, and soy food consumption.
* Participants will return the surveys to the researchers in the stamped envelope provided with the questionnaire....

DETAILED DESCRIPTION:
We propose a follow-up study of women who participated in the North Carolina Early Pregnancy Study (EPS) in 1982-1986. Women enrolled in the study after discontinuing birth control and were followed for the occurrence of a pregnancy. Participants completed daily diaries and collected first morning urine specimens which allowed the identification of menstrual cycles. Thus each woman s time to pregnancy was prospectively measured. We intend to trace the women and ask them to complete a questionnaire that includes their recall of their time to pregnancy during the study. This will allow us to address two major questions, one regarding the recall of time-to-pregnancy, and the other regarding the natural length of gestation. In addition, we will investigate associations of bisphenal A (BPA), phthalate metabolites, 2,4- and 2,5-dichlorophenols, Triclosan, benzophenone-3, and methyl-, propyl- and butyl-parabens with reproductive outcomes. This is described in a separate section at the end of this protocol because it does not involve recontacting participants, only assay of stored urine samples for purposes within the goals of the original study.

1. Recall of time-to-pregnancy

   Time to pregnancy is a commonly studied estimate of fecundability. This outcome has been used to study the reproductive effects of environmental toxins, cigarette smoking, obesity and numerous other exposures. Prospective studies of time to pregnancy require enrollment of women who are just starting to attempt pregnancy and following them until a pregnancy is conceived. This type of study can be time-consuming and costly. It is also difficult to identify a population of women who are just beginning to attempt pregnancy. A more efficient design is to ask women to recall their time to pregnancy. This design is limited however, as it is unknown how well women can recall their time to pregnancy. Only two studies have examined this question in a population with both prospective and retrospectively recalled time to pregnancy. One of the studies involved women from the Netherlands, the recall period was short (3-20 months), and only part of the woman s time to pregnancy was prospectively observed. The second study had a longer recall period (1-10 years) but included only 43 women.
2. Length of gestation

Gestational length is the time from conception to delivery. The EPS has very good data on the first data point, and we know date of delivery. However, our data on delivery is limited by the fact that we do not know which deliveries were induced and which were the product of natural onset of labor and delivery. We plan to collect this information from the mothers. Such information will not only allow us to consider the natural variability in gestational age (a measure that does not exist at present) but also to estimate associations between events in very early pregnancy and the subsequent duration of pregnancy. The EPS has detailed measurements of the time from ovulation to implantation, the rate of increase in human chorionic gonadotropin and corpus luteum rescue. To our knowledge, these early pregnancy characteristics have not been investigated for associations with length of gestation.

ELIGIBILITY:
* INCLUSION AND EXCLUSION CRITERIA:

This study is a follow-up study of women who participated in the NIEHS EPS. All of the women who participated in that study are eligible for this follow-up.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who participated in the 1982-1986 North Carolina Early Pregnancy Study (EPS)
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2010-05-05 (Actual); Primary Completion 2011-09-02 (Actual); Study Completion 2017-02-24 (Actual)

PRIMARY OUTCOMES:
Gestation Length | Retrospective recall
  Recall of time to pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Marie Z Jukic, Ph.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- NIEHS, Research Triangle Park, Research Triangle Park, North Carolina, United States